CLINICAL TRIAL: NCT00278057
Title: PHASE 4 STUDY OT THE EFFECT OF GLUCOSE ADDED TO THE DIALYSIS FLUID ON BLOOD PRESSURE, BLOOD GLUCOSE AND QUALITY OF LIFE IN HEMODIALYSIS PATIENTS.
Brief Title: STUDY OF GLUCOSE IN DIALYSIS WATER WITH REGARD TO BLOOD PRESSURE AND QUALITY OF LIFE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Other Study IDs: MED. RES. HOS.2003.01
Record Dates: First submitted 2006-01-16; First posted 2006-01-18 (Estimated); Last update posted 2006-01-18 (Estimated); Status verified 2006-01

CONDITIONS: Hemodialysis
Keywords: Blood pressure;; chronic renal failure;; diabetes mellitus;; dialysis fluid; glucose;; hemodialysis;; hypertension;; uremia.
MeSH Terms: conditions — Kidney Failure, Chronic; Diabetes Mellitus; Hypertension; Uremia | interventions — Glucose

INTERVENTIONS:
Drug: dialysisis with and without glucose in the dialysis

SUMMARY:
We wanted to test the hypotheses that blood pressure level was lower, that the variability of blood pressure and blood glucose was reduced, and that quality of life was improved when glucose was added to the dialysis fluid.

DETAILED DESCRIPTION:
The purpose of the study was to determine the effect of glucose added to the dialysis fluid on 1.blood pressure and variation in blood pressure, 2.blood glucose and variation in blood glucose, and 3.quality of life in patients treated with chronic maintenance hemodialysis in a randomized, placebo-controlled, unblinded cross-over study.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18 years, both men and women, and hemodialysis treatment for more than three months

Exclusion Criteria:

* treatment with hemodiafiltration, change to another dialysis modality, renal transplantation, alcohol abuse defined as more than 21 drinks a week for men and more than 14 drinks a week for women, and unwillingness to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55
Dates: Start 2003-05; Study Completion 2003-05

CONTACTS AND LOCATIONS:
Overall Officials: Erling B Pedersen, Professor, Study Chair — Holstebro Hospital, 7500 Holstebro, Denmark
Locations (1):
- Department of Medicine, Holstebro Hospital, Holstebro, Denmark